CLINICAL TRIAL: NCT01826006
Title: A Randomized Comparison of Excimer LASER vs Manual Thrombus Aspiration for the Prevention of No-reflow During Primary Percutaneous Coronary Intervention of St-elevation Myocardial Infarction(LASER-AMI Study)
Brief Title: THE LASER-AMI STUDY - Excimer Laser Versus Manual Thrombus Aspiration in Acute Myocardial Infarction
Acronym: LASER-AMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, GIANPAOLO NICCOLI, Dott. Prof., Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LASER-AMI P/915/CE/2012; LASER-AMI P/915/CE/2012
Record Dates: First submitted 2013-03-28; First posted 2013-04-08 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; No-reflow; Primary PCI; Coronary no-reflow phenomenon; Primary percoutaneous coronary intervention (primary PCI)
MeSH Terms: conditions — Myocardial Infarction | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Excimer laser (Active Comparator): After wire crossing, Excimer Laser will be performed. Consequently, intracoronary adenosine will be selectively administered through the guiding catheter.
  Interventions: Device: Excimer laser
- Manual Thrombus Aspiration (Active Comparator): After wire crossing, thrombus aspiration will be performed. The device will removed outside the body, flushed with saline and subsequently reintroduced in the culprit vessel beyond the occlusion site and intracoronary adenosine will be selectively administered.
  Interventions: Device: Manual Thrombus Aspiration

INTERVENTIONS:
Device: Excimer laser
  Arms: Excimer laser
Device: Manual Thrombus Aspiration
  Arms: Manual Thrombus Aspiration

SUMMARY:
The occurrence of no-reflow phenomenon after recanalization of the infarct related artery in acute myocardial infarction is described in up to 40% of cases. This event is associated with a worse prognosis at follow up and an unfavourable left ventricular remodelling. Two main pathogenetic mechanisms cause no-reflow: distal embolization, ischemia-reperfusion injury and individual susceptibility. In such a context, Excimer Laser (EL) may play an important role in order to reduce the rate of microvascular obstruction.

Thus, in this randomized study we will assess the effect of EL versus Manual Thrombus Aspiration for ST elevation MI using ST segment resolution on standard 12 leads ECG as primary endpoint of myocardial reperfusion.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is the leading cause of death in developed countries. In patients with AMI, prompt reopening of an occluded coronary artery is the main goal of reperfusion therapies in order to restore normal blood flow to the myocardium, thus preventing left ventricular (LV) adverse remodelling and occurrence of heart failure. Primary percutaneous coronary intervention (PPCI) represents the pivotal step in the current management of ST-segment elevation myocardial infarction (STEMI) (1). Yet, in a sizable proportion of patients, PPCI achieves epicardial coronary artery reperfusion but not myocardial reperfusion, a condition known as no-reflow (2), that increases the extent of myocardial damage. The proportion of patients who get optimal myocardial reperfusion, among those without cardiogenic shock undergoing PPCI, is about 35% (3). Thus, the prevalence of no-reflow remains extremely high. Furthermore, a series of consistent data has clearly shown that no-reflow has a strong negative impact on outcome, negating the potential benefit of PPCI (4-10). Indeed, as compared to patients without no-reflow, patients with no-reflow exhibit a higher prevalence of: 1) early post-infarction complications (arrhythmias, pericardial effusion, cardiac tamponade, early congestive heart failure); 2) LV adverse remodelling; 3) late re-hospitalizations for heart failure; 4) mortality. In man, no-reflow is caused by the variable combination of four pathogenetic mechanisms: 1) distal atherothrombotic embolization, 2) ischemic injury, 3) reperfusion injury, 4) susceptibility of coronary microcirculation to injury (3). As a consequence, appropriately designed strategies to prevent or to treat, at the right time, each of these components are expected to reduce the final number of patients with no-reflow. Manual thrombus aspiration (MTA) has been clearly shown to improve microvascular perfusion and survival in STEMI patients treated by PPCI (9,10). Accordingly, in current guidelines of the European Society of Cardiology (ESC), MTA is a 2a recommendation (1). Yet, complete ST-segment resolution (defined as >70%) is obtained in only about 50% of patients (3,6), thus suggesting that microvascular perfusion may be further improved. In such a context, Excimer laser (EL) may play an important role in order to reduce the rate of microvascular obstruction. Coronary lasers are devices emitting electromagnetic energy which, upon absorption within the atherosclerotic plaque, can debulk the target tissue (11-12). Over the past decade, a second generation of pulsed-wave lasers was introduced (13). These devices combine a brief pulse duration of light emission with a long pause interval, thus ensuring prevention of thermal injury and adverse effect on the arterial wall to be laser. The pulsed wave EL (308 nm, ultraviolet wavelength, in the UVB region of the spectrum) is an FDA and EMEA approved device for treatment of atherosclerotic coronary lesions considered "non ideal" for standard balloon angioplasty (14-16). Furthermore, continuous saline flush of saline during laser advancement has allowed to further reduce heat generation and tissue damage. Taken together device improvement and technical advancement have allowed to lower procedural complication rate and to confirm in published registries the safety of the EL assisted angioplasty (17-18). In the setting of thrombotic lesion, EL has the potential to vaporize thrombotic and plaque material, leading to particles smaller than the size of erythrocytes unlikely to plug the microcirculation (19-20), and inhibits platelet aggregation, by inducing platelets stunning (21). Furthermore, laser is able to debulk underlying thrombogenic plaque thus limiting its thrombogenicity (22). EL has been used in the setting of STEMI within registries (23-26) and in a small randomized trial vs balloon assisted PPCI (27), showing a very low rate of myocardial no-reflow, as assessed by angiography (around 5%) and electrocardiography (around 35%). These studies, however, were limited by the small sample size and for most of them by the non-randomized design. Thus, a randomized study of EL assisted PPCI has become necessary in order to evaluate the efficacy of this mechanical strategy for STEMI patients. As MTA-assisted PPCI is nowadays the recommended approach by current guidelines, the effectiveness of EL-assisted PPCI should be evaluated against MTA-assisted PPCI. The goal of this trial, which will be carried out in patients with STEMI undergoing PPCI, is to assess the superiority of EL-assisted vs MTA-assisted PPCI, having as primary end-point the rate of 90-min ST segment resolution>70% and as secondary end-points the rate of angiographic no-reflow, defined as TIMI flow3 and MBG >=2 (28), the evaluation of infarct size, as assessed by the area under the curve of cardiac markers (29) and the rate of adverse remodelling as assessed by echocardiography at 6 months follow-up

Description of LASER-AMI trial

Study design

LASER-AMI is a randomized, open-label, blind-examination (PROBE), active controlled, multinational clinical trial. Patients undergoing PPCI will be randomly assigned to 1 of 2 interventional strategies of reperfusion: MTA-assisted PPCI alone or EL-assisted PPCI alone.

Study protocol and procedure

The informed consent will be signed before angiography. The randomization process will start after the completion of diagnostic angiography and patients will be allocated to one of the following two arms: MTA-assisted PPCI alone; or EL-assisted PPCI alone. A consecutively numbered and sealed envelope will be opened to have knowledge of the randomization arm. Each enrolling center will receive from the promoting center an exact number of numbered envelopes to use for the randomization.

The interventional procedure will be carried out according to usual site's local protocol. The choice of vascular access and stent type will be left to operator discretion. All patients will receive aspirin per os (150-325 mg), clopidogrel (600 mg) or prasugrel or ticagrelor in the emergency department. Anticoagulant therapy in the catheterization laboratory will be left to the operator's choice according to recent ESC guidelines (1); GP IIb/IIIa inhibitors will be considered for bailout therapy if there is angiographic evidence of massive thrombus, slow or no-reﬂow or a thrombotic complication. After identification of culprit vessel and crossing the lesion by the guidewire, vessel recanalization will start by using either MTA or EL, according to randomization (see appendix 1 about advices for ELCA use). The choice of the MTA devices will be left to each site's usual availability. Complications related to either ELCA or MTA will be recorded (perforation, dissection) as well as failure to restore antegrade flow and lack of crossing culprit stenosis. The use of balloon after MTA or EL is left to operator discretion, even if direct stenting is recommended. In all patients, after MTA or ELCA, intracoronary adenosine (120 µg as fast bolus followed by 2 mg given in 33cc of saline in 2 minutes as slow bolus) will be administered.

Vessel recanalization will be completed by coronary stenting. Postdilatation of the stent is left to the operator's discretion, although stent overexpansion is not recommended in order to reduce the risk for no-reflow.

Angiographic and electrocardiography analysis

Angiographic analysis will be performed off-line by the angio core lab (IsMeTT, Palermo, Italy) and will include: quantitative coronary angiography (31), TIMI flow (32), corrected TIMI frame count (33), MBG (34), combined evaluation of TIMI flow and MBG (27), thrombus score (35), and Rentrop collateral grading (36). Angiographic no-reflow will be defined as a final TIMI flow of < 2 or final TIMI flow 3 with a MBG 0/1 (3,27). These parameters will be assessed according to validated methods (31-36).

At 90 minutes after the end of the procedure a 12 leads ECG will be recorded for the analysis of ST-segment resolution as compared to admission ECG. Complete ST-segment resolution will be defined as >70% of ST-segment as compared to baseline in both single lead showing maximum ST-elevation on admission and on the sum of leads showing ST-elevation on admission (37,38) Baseline ECG will be also assessed off-line for number of Q waves and terminal distorsion of QRS (39).

ECG analysis will be performed offline by an ECG core lab (Clinica di Cardiologia, UNIVPM, Ancona, Italy).

Echocardiographic protocol

At day 3 to 5 and at 6-month after the index procedure all patients will undergo comprehensive 2D transthoracic echocardiography examination at rest. End-systolic (LVESV) and end-diastolic volumes (LVEDV), LV ejection fraction (LVEF), presence and degree of mitral insufficiency and wall motion score index (each segment scored from 1= normal/ hyperkinetic, to 4 = dyskinetic, in a 16 segment model of the left ventricle) will be calculated following the recommendations of the American Society of Echocardiography (40). LV volumes and ejection fraction will be measured by modified biplane Simpson's method, and adjusted for body surface area. LV remodeling will be defined as an increase in end-diastolic volume > 20% at 6 months after AMI as compared to in-hospital examination (7).

Serious Adverse Events

Serious adverse events will be recorded and defined as any untoward medical occurrence that results in cardiac death, vascular death, death, re-infarction, target lesion revascularization, target vessel revascularization, or stent thrombosis. They will be communicated to the Safety Board within 24hours from their occurrence.

Blood sampling

Blood samples will be collected before the PCI and at 4, 8, 12, 24, 36, 48, and 72 h after the procedure to measure creatine kinase-myocardial band (CK-MB) (mass), troponin-T (mass), and hemoglobin levels.

Clinical follow-up

The incidence of cardiac death, myocardial infarction, target lesion revascularization and heart failure requiring hospitalization will be assessed at 6 months by interview and clinical check and at 1 year by telephone contact. In line with protocol, interviewers and examiners will not know which drug was administrated at the time of procedure. The accumulation of such end-points will be defined as major adverse cardiac events (MACEs).

Study end-point

The end-point of the study is the comparison of the rate of ST-segment resolution at 90 minutes post PPCI between patients randomized to MTA-assisted PPCI and EL-assisted PPCI. Thus, the study will test whether EL-assisted PPCI is superior to MTA-assisted PPCI in reducing of the incidence of electrocardiographic no-flow after performing PPCI.

Secondary endpoints are: a) angiographic no-reflow defined as a TIMI flow ≤2 or a TIMI flow 3 with a MBG 0/1; b) LVESV, LVEDV, LVEF, and WMSI assessed by in-hospital and 6 months echocardiography; c) infarct size, defined as CK-MB and troponin-I area under the curve; d) MACEs rate in the two groups at 6 and 1 year follow-up.

Power calculation

LASER-AMI is a randomized, open-label clinical trial, in which patients will be randomly assigned to 1 of 2 interventional strategies (MTA-assisted PPCI; or EL-assisted PPCI). The primary objective of LASER-AMI trial is to test the superiority of EL-assisted PPCI vs MTA-assisted PPCI based on the rate of post-procedural STR>70% after PPCI. The study sample size was powered to demonstrate a significant difference in the primary end point of rate STR >70%, which was around 56% in a previous trial of PPCI with MTA only (10). Starting from such figures and thus assuming an 76% event rate in the control group with an absolute 20% decrease in the experimental group, we calculated that 194 patients (97 per group) had to be enrolled to have an alpha error of 0.05 and a power of 0.80 in a prospective 1:1 randomized study.

Statistical analysis

All analyses will be planned and conducted according to the intention-to-treat principle, as this approach minimizes the risk of selection bias and alpha error. Continuous variables (presented as mean ± standard deviation) will be compared by the Student t test for normally distributed variables and by the Wilcoxon test for nonnormally distributed variables. Chi-square tests will be used to compare discrete variables (reported as raw numbers [%]). Odds ratios (OR) with 95% confidence intervals (CI) will be calculated to compare event rates in the EL-assisted PPCI group versus those observed in the MTA-assisted PPCI group (considered as the control group). A multivariable logistic regression analysis will be also performed to further assess and confirm the independent predictive value of randomization to EL-assisted PPCI for the achievement of STR>70% (cut-off for entry 0.05, cut-off for removal 0.10). Moreover, infarct size assessment will be perfomed, defined as CK-MB and troponin-I area under the curve, calculated by the linear trapezoidal method (29). If baseline or 72-h values are missing, the value will be set to 0, whereas missing intermediate values will be substituted by linear interpolation. For patients dying in the first 72 h after enrollment, the area under the curve will be set as the largest area under the curve recorded in the study (29). Analyses will be carried out using SPSS for Windows 11.0 (SPSS Inc., Chicago, Illinois). Statistical significance will be defined by two-tailed p < 0.05.

In addition, prespecified subgroup analyses by means of multiple logistic regression or multiple linear regression, as appropriate, will be performed according to the following variables: age class, sex, diabetes, anterior myocardial infarction, total ischemic time cutoff, pre-infarction angina, baseline angiographic thrombus score, baseline TIMI flow, number of diseased vessels.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms of MI less than 12 hours prior to enrolment;
* ST-segment elevation of at least 2 mm in two or more contiguous leads;
* Vessel and lesion amenable to both coronary laser and manual trhombus aspiration (lack of marked vessel/lesion tortuosity or calcification; reference vessel diameter >2.5 mm in diameter);
* Written informed consent.

Exclusion Criteria:

* Rescue angioplasty after failed thrombolysis;
* Stent thrombosis;
* Culprit lesion located in a bypass graft or in the left main trunk;
* Cardiogenic shock;
* Young age (< 18 years);
* Severe renal failure (creatinine clearance ≤30 ml/min);
* Concomitant disease resulting in a life expectancy of less than 6 months;
* Pregnancy;
* Contraindications to contrast agents not manageable medically, or to study medications, including aspirin, clopidogrel, ticlopidine and heparin;
* Left bundle branch block, paced rhythm, frequent ventricular ectopy, pre-excitation or other ECG abnormalities interfering with the analysis of ST-segment resolution;
* Markedly depressed LV function (LVEF <30%); Culprit lesion cannot be identified;
* Severe left main or triple vessel disease requiring CABG during the index hospitalization;
* Patients already involved in other ongoing trials;
* Patients unable or unwilling to give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Medicina Cardiovascolare, Rome, Italy

REFERENCES:
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Rezkalla SH, Kloner RA. No-reflow phenomenon. Circulation. 2002 Feb 5;105(5):656-62. doi: 10.1161/hc0502.102867. No abstract available. PMID 11827935
- [Background] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92. doi: 10.1016/j.jacc.2009.03.054. PMID 19608025
- [Background] Brosh D, Assali AR, Mager A, Porter A, Hasdai D, Teplitsky I, Rechavia E, Fuchs S, Battler A, Kornowski R. Effect of no-reflow during primary percutaneous coronary intervention for acute myocardial infarction on six-month mortality. Am J Cardiol. 2007 Feb 15;99(4):442-5. doi: 10.1016/j.amjcard.2006.08.054. Epub 2006 Dec 20. PMID 17293180
- [Background] Henriques JP, Zijlstra F, van 't Hof AW, de Boer MJ, Dambrink JH, Gosselink M, Hoorntje JC, Suryapranata H. Angiographic assessment of reperfusion in acute myocardial infarction by myocardial blush grade. Circulation. 2003 Apr 29;107(16):2115-9. doi: 10.1161/01.CIR.0000065221.06430.ED. Epub 2003 Apr 14. PMID 12695301
- [Background] McLaughlin MG, Stone GW, Aymong E, Gardner G, Mehran R, Lansky AJ, Grines CL, Tcheng JE, Cox DA, Stuckey T, Garcia E, Guagliumi G, Turco M, Josephson ME, Zimetbaum P; Controlled Abciximab and Device Investigation to Lower Late Angioplasty Complications trial. Prognostic utility of comparative methods for assessment of ST-segment resolution after primary angioplasty for acute myocardial infarction: the Controlled Abciximab and Device Investigation to Lower Late Angioplasty Complications (CADILLAC) trial. J Am Coll Cardiol. 2004 Sep 15;44(6):1215-23. doi: 10.1016/j.jacc.2004.06.053. PMID 15364322
- [Background] Bolognese L, Carrabba N, Parodi G, Santoro GM, Buonamici P, Cerisano G, Antoniucci D. Impact of microvascular dysfunction on left ventricular remodeling and long-term clinical outcome after primary coronary angioplasty for acute myocardial infarction. Circulation. 2004 Mar 9;109(9):1121-6. doi: 10.1161/01.CIR.0000118496.44135.A7. Epub 2004 Feb 16. PMID 14967718
- [Background] Galiuto L, Garramone B, Scara A, Rebuzzi AG, Crea F, La Torre G, Funaro S, Madonna M, Fedele F, Agati L; AMICI Investigators. The extent of microvascular damage during myocardial contrast echocardiography is superior to other known indexes of post-infarct reperfusion in predicting left ventricular remodeling: results of the multicenter AMICI study. J Am Coll Cardiol. 2008 Feb 5;51(5):552-9. doi: 10.1016/j.jacc.2007.09.051. PMID 18237684
- [Background] Burzotta F, Trani C, Romagnoli E, Mazzari MA, Rebuzzi AG, De Vita M, Garramone B, Giannico F, Niccoli G, Biondi-Zoccai GG, Schiavoni G, Mongiardo R, Crea F. Manual thrombus-aspiration improves myocardial reperfusion: the randomized evaluation of the effect of mechanical reduction of distal embolization by thrombus-aspiration in primary and rescue angioplasty (REMEDIA) trial. J Am Coll Cardiol. 2005 Jul 19;46(2):371-6. doi: 10.1016/j.jacc.2005.04.057. PMID 16022970
- [Background] Svilaas T, Vlaar PJ, van der Horst IC, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Thrombus aspiration during primary percutaneous coronary intervention. N Engl J Med. 2008 Feb 7;358(6):557-67. doi: 10.1056/NEJMoa0706416. PMID 18256391
- [Background] Grundfest WS, Segalowitz J, Laudenslager JB, et al. The physical and biological basis for laser angioplasty. In: Litvack F, editor. Coronary laser angioplasty. Oxford: Blackwell Scientific Publications, 1992:5-12
- [Background] van Leeuwen TG, Borst C. Fundamental laser-tissue interactions. Semin Interv Cardiol. 1996 Jun;1(2):121-8. PMID 9552502
- [Background] Haase KK, Rose C, Duda S, Baumbach A, Oberhoff M, Anthanasiadis A, Karsch KR. Perspectives of coronary excimer laser angioplasty: multiplexing, saline flushing, and acoustic ablation control. Lasers Surg Med. 1997;21(1):72-8. doi: 10.1002/(sici)1096-9101(1997)21:13.0.co;2-b. PMID 9228643
- [Background] Linsker R, Srinivasan R, Wynne JJ, Alonso DR. Far-ultraviolet laser ablation of atherosclerotic lesions. Lasers Surg Med. 1984;4(2):201-6. doi: 10.1002/lsm.1900040212. PMID 6472033
- [Background] Grundfest WS, Litvack F, Forrester JS, Goldenberg T, Swan HJ, Morgenstern L, Fishbein M, McDermid IS, Rider DM, Pacala TJ, et al. Laser ablation of human atherosclerotic plaque without adjacent tissue injury. J Am Coll Cardiol. 1985 Apr;5(4):929-33. doi: 10.1016/s0735-1097(85)80435-6. PMID 3838324
- [Background] Isner JM, Donaldson RF, Deckelbaum LI, Clarke RH, Laliberte SM, Ucci AA, Salem DN, Konstam MA. The excimer laser: gross, light microscopic and ultrastructural analysis of potential advantages for use in laser therapy of cardiovascular disease. J Am Coll Cardiol. 1985 Nov;6(5):1102-9. doi: 10.1016/s0735-1097(85)80316-8. PMID 4045033
- [Background] Bittl JA, Sanborn TA. Excimer laser-facilitated coronary angioplasty. Relative risk analysis of acute and follow-up results in 200 patients. Circulation. 1992 Jul;86(1):71-80. doi: 10.1161/01.cir.86.1.71. PMID 1617792
- [Background] Margolis JR, Mehta S. Excimer laser coronary angioplasty. Am J Cardiol. 1992 May 7;69(15):3F-11F. doi: 10.1016/0002-9149(92)91176-5. PMID 1621649
- [Background] Topaz O, Shah R, Mohanty PK, McQueen RA, Janin Y, Bernardo NL. Application of excimer laser angioplasty in acute myocardial infarction. Lasers Surg Med. 2001;29(2):185-92. doi: 10.1002/lsm.1108. PMID 11553909
- [Background] Topaz O, Bernardo NL, Shah R, McQueen RH, Desai P, Janin Y, Lansky AJ, Carr ME. Effectiveness of excimer laser coronary angioplasty in acute myocardial infarction or in unstable angina pectoris. Am J Cardiol. 2001 Apr 1;87(7):849-55. doi: 10.1016/s0002-9149(00)01525-3. PMID 11274939
- [Background] Topaz O, Minisi AJ, Bernardo NL, McPherson RA, Martin E, Carr SL, Carr ME Jr. Alterations of platelet aggregation kinetics with ultraviolet laser emission: the "stunned platelet" phenomenon. Thromb Haemost. 2001 Oct;86(4):1087-93. PMID 11686328
- [Background] Ferrante G, Cosentino N, Conte M, et al. Rescue excimer laser coronary angioplasty after manual thrombus aspiration failure in acute ST-elevation myocardial infarction. Il Giornale Italiano di Cardiologia Invasiva 2009,2:9-12
- [Background] Topaz O, Ebersole D, Das T, Alderman EL, Madyoon H, Vora K, Baker JD, Hilton D, Dahm JB; CARMEL multicenter trial. Excimer laser angioplasty in acute myocardial infarction (the CARMEL multicenter trial). Am J Cardiol. 2004 Mar 15;93(6):694-701. doi: 10.1016/j.amjcard.2003.11.050. PMID 15019871
- [Background] Dahm JB, Ebersole D, Das T, Madyhoon H, Vora K, Baker J, Hilton D, Topaz O. Prevention of distal embolization and no-reflow in patients with acute myocardial infarction and total occlusion in the infarct-related vessel: a subgroup analysis of the cohort of acute revascularization in myocardial infarction with excimer laser-CARMEL multicenter study. Catheter Cardiovasc Interv. 2005 Jan;64(1):67-74. doi: 10.1002/ccd.20239. PMID 15619312
- [Background] Dave RM. Excimer laser in acute myocardial infarction: first report of the Extended FAMILI Study. TCT, 2006
- [Background] Ambrosini V, Cioppa A, Salemme L, Tesorio T, Sorropago G, Popusoi G, Stabile E, Medolla A, Cangella F, Agrusta M, Picano E, Rubino P. Excimer laser in acute myocardial infarction: single centre experience on 66 patients. Int J Cardiol. 2008 Jun 23;127(1):98-102. doi: 10.1016/j.ijcard.2007.10.060. Epub 2008 Feb 15. PMID 18280596
- [Background] Dorr M, Vogelgesang D, Hummel A, Staudt A, Robinson DM, Felix SB, Dahm JB. Excimer laser thrombus elimination for prevention of distal embolization and no-reflow in patients with acute ST elevation myocardial infarction: results from the randomized LaserAMI study. Int J Cardiol. 2007 Mar 2;116(1):20-6. doi: 10.1016/j.ijcard.2006.03.024. Epub 2006 Aug 7. PMID 16891005
- [Background] Gibson CM, Murphy SA, Morrow DA, Aroesty JM, Gibbons RJ, Gourlay SG, Barron HV, Giugliano RP, Antman EM, Braunwald E. Angiographic perfusion score: an angiographic variable that integrates both epicardial and tissue level perfusion before and after facilitated percutaneous coronary intervention in acute myocardial infarction. Am Heart J. 2004 Aug;148(2):336-40. doi: 10.1016/j.ahj.2003.12.044. PMID 15309006
- [Background] Patti G, Barczi G, Orlic D, Mangiacapra F, Colonna G, Pasceri V, Barbato E, Merkely B, Edes I, Ostojic M, Wijns W, Di Sciascio G. Outcome comparison of 600- and 300-mg loading doses of clopidogrel in patients undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: results from the ARMYDA-6 MI (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty-Myocardial Infarction) randomized study. J Am Coll Cardiol. 2011 Oct 4;58(15):1592-9. doi: 10.1016/j.jacc.2011.06.044. PMID 21958886
- [Background] Perazzolo Marra M, Lima JA, Iliceto S. MRI in acute myocardial infarction. Eur Heart J. 2011 Feb;32(3):284-93. doi: 10.1093/eurheartj/ehq409. Epub 2010 Nov 25. PMID 21112897
- [Background] Hermiller JB, Cusma JT, Spero LA, Fortin DF, Harding MB, Bashore TM. Quantitative and qualitative coronary angiographic analysis: review of methods, utility, and limitations. Cathet Cardiovasc Diagn. 1992 Feb;25(2):110-31. doi: 10.1002/ccd.1810250207. PMID 1544153
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Gibson CM, Cannon CP, Daley WL, Dodge JT Jr, Alexander B Jr, Marble SJ, McCabe CH, Raymond L, Fortin T, Poole WK, Braunwald E. TIMI frame count: a quantitative method of assessing coronary artery flow. Circulation. 1996 Mar 1;93(5):879-88. doi: 10.1161/01.cir.93.5.879. PMID 8598078
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Yip HK, Chen MC, Chang HW, Hang CL, Hsieh YK, Fang CY, Wu CJ. Angiographic morphologic features of infarct-related arteries and timely reperfusion in acute myocardial infarction: predictors of slow-flow and no-reflow phenomenon. Chest. 2002 Oct;122(4):1322-32. doi: 10.1378/chest.122.4.1322. PMID 12377860
- [Background] Rentrop KP, Cohen M, Blanke H, Phillips RA. Changes in collateral channel filling immediately after controlled coronary artery occlusion by an angioplasty balloon in human subjects. J Am Coll Cardiol. 1985 Mar;5(3):587-92. doi: 10.1016/s0735-1097(85)80380-6. PMID 3156171
- [Background] Schroder R, Dissmann R, Bruggemann T, Wegscheider K, Linderer T, Tebbe U, Neuhaus KL. Extent of early ST segment elevation resolution: a simple but strong predictor of outcome in patients with acute myocardial infarction. J Am Coll Cardiol. 1994 Aug;24(2):384-91. doi: 10.1016/0735-1097(94)90292-5. PMID 8034872
- [Background] van 't Hof AW, Liem A, de Boer MJ, Zijlstra F. Clinical value of 12-lead electrocardiogram after successful reperfusion therapy for acute myocardial infarction. Zwolle Myocardial infarction Study Group. Lancet. 1997 Aug 30;350(9078):615-9. doi: 10.1016/s0140-6736(96)07120-6. PMID 9288043
- [Background] Lee CW, Hong MK, Yang HS, Choi SW, Kim JJ, Park SW, Park SJ. Determinants and prognostic implications of terminal QRS complex distortion in patients treated with primary angioplasty for acute myocardial infarction. Am J Cardiol. 2001 Aug 1;88(3):210-3. doi: 10.1016/s0002-9149(01)01627-7. PMID 11472695
- [Background] Schiller NB, Shah PM, Crawford M, DeMaria A, Devereux R, Feigenbaum H, Gutgesell H, Reichek N, Sahn D, Schnittger I, et al. Recommendations for quantitation of the left ventricle by two-dimensional echocardiography. American Society of Echocardiography Committee on Standards, Subcommittee on Quantitation of Two-Dimensional Echocardiograms. J Am Soc Echocardiogr. 1989 Sep-Oct;2(5):358-67. doi: 10.1016/s0894-7317(89)80014-8. PMID 2698218